CLINICAL TRIAL: NCT07371676
Title: Acute Effects of Post-Exercise Vagus Nerve Stimulation on the Autonomic Nervous System and Recovery in Healthy Young Adults
Brief Title: Effects of Vagus Nerve Stimulation on the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19.04.2024/05
Record Dates: First submitted 2025-12-29; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Auricular Vagus Nerve Stimulation; Transcutaneous; Recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve stimulation group (Experimental)
  Interventions: Device: Stimulation
- Control Group (No Intervention)

INTERVENTIONS:
Device: Stimulation — Recovery in athletes through vagus nerve stimulation
  Arms: Vagus nerve stimulation group

SUMMARY:
The aim of this study is to determine the effect of vagus nerve stimulation, applied after running exercise, on recovery and fatigue in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy between the ages of 18-35
* Volunteering to participate in the study
* Signing the voluntary consent form
* Being in the inactive category according to the International Physical Activity Questionnaire

Exclusion Criteria:

* Having a regular exercise habit
* Being in the very minimally active or active category according to the International Physical Activity Survey
* Presence of any chronic disease and medication use for this condition
* History and treatment of current respiratory system disease
* History and treatment of current cardiac system disease
* History and treatment of current hearing system disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the autonomic nervous system. | Periprocedural
  Using heart rate variability (HRV) measurements recorded

SECONDARY OUTCOMES:
Lactic acid concentrate indicator | Periprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gelisim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim AY, Marduy A, de Melo PS, Gianlorenco AC, Kim CK, Choi H, Song JJ, Fregni F. Safety of transcutaneous auricular vagus nerve stimulation (taVNS): a systematic review and meta-analysis. Sci Rep. 2022 Dec 21;12(1):22055. doi: 10.1038/s41598-022-25864-1. PMID 36543841
- [Background] Ackland GL, Patel ABU, Miller S, Gutierrez Del Arroyo A, Thirugnanasambanthar J, Ravindran JI, Schroth J, Boot J, Caton L, Mein CA, Abbott TEF, Gourine AV. Non-invasive vagus nerve stimulation and exercise capacity in healthy volunteers: a randomized trial. Eur Heart J. 2025 May 2;46(17):1634-1644. doi: 10.1093/eurheartj/ehaf037. PMID 39969124
- [Background] Hatik SH, Arslan M, Demirbilek O, Ozden AV. The effect of transcutaneous auricular vagus nerve stimulation on cycling ergometry and recovery in healthy young individuals. Brain Behav. 2023 Dec;13(12):e3332. doi: 10.1002/brb3.3332. Epub 2023 Nov 16. PMID 37974551